CLINICAL TRIAL: NCT00640198
Title: A 24-Week Pilot, Double-Blind, Randomized, Parallel, Placebo-Controlled Study of Memantine and Constraint-Induced Language Therapy in Chronic Poststroke Aphasia:Correlation With Cognitive Evoked Potentials During Recovery.
Brief Title: Memantine and Intensive Speech-Language Therapy in Aphasia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gabinete Berthier y Martínez (Other)
Collaborators: H. Lundbeck A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M-10830; Gabinete Berthier y Martínez.; Lundbeck, Spain, S.A.
Record Dates: First submitted 2008-03-17; First posted 2008-03-21 (Estimated); Last update posted 2008-03-21 (Estimated); Status verified 2008-03

CONDITIONS: Aphasia; Stroke
Keywords: Aphasia; Memantine; Constraint-induced language therapy; Event-related potentials
MeSH Terms: conditions — Aphasia; Stroke | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 Memantine (Active Comparator): Patients included in this group will receive memantine alone followed by memantine combined with intensive speech-language therapy.
  Interventions: Drug: memantine; Behavioral: constraint-induced language therapy (CIAT)
- Group 2 (Placebo Comparator): Patients included in this group will receive placebo alone followed by memantine combined with intensive speech-language therapy.
  Interventions: Behavioral: constraint-induced language therapy (CIAT); Drug: placebo

INTERVENTIONS:
Drug: memantine — Memantine was titrated in 5-mg weekly increments as recommended,from a starting dose of 5 mg/day to 20 mg/day. After the 3-week up-titration phase all patients received a fixed dose of either memantine (10 mg) or placebo twice daily without CIAT during the next 3 months (week 16). During the next 2 weeks (weeks 16-18), the drug treatment was combined with CIAT. This phase of combined treatment was followed by a 2-week period (weeks 18-20) where patients received memantine or placebo treatment alone and, finally, by a 4-week period of drug withdrawal (weeks 20-24)
  Other Names: Ebixa, Namenda
  Arms: Group 1 Memantine
Behavioral: constraint-induced language therapy (CIAT) — CIAT is an intensive form of language-action therapy for aphasia performed in a small group setting. In a therapeutic game context, participants had to request objects or cards from each other and understand requests made by others. Feedback of communicative success was regularly given, along with guidance, help and reinforcement. Gesturing replacing verbal language was discouraged although gestures accompanying speech were allowed. Difficulty levels were adjusted to the patients´ communicative abilities by choosing language materials and actions and reinforcement was administered taking into account each patient´s level of performance. Communication rules were introduced by shaping and modelling. Each patient received 30 hours of therapy.
  Other Names: Intensive language-action therapy
Drug: memantine — Memantine was titrated in 5-mg weekly increments as recommended, from a starting dose of 5 mg/day to 20 mg/day. After the 3-week up-titration phase all patients received a fixed dose of either memantine (10 mg) or placebo twice daily without CIAT during the next 3 months (week 16). During the next 2 weeks (weeks 16-18), the drug treatment was combined with CIAT. This phase of combined treatment was followed by a 2-week period (weeks 18-20) where patients received memantine or placebo treatment alone and, finally, by a 4-week period of drug withdrawal (weeks 20-24).
  Other Names: Ebixa, Namenda
  Arms: Group 1 Memantine
Drug: placebo — Placebo
  Arms: Group 2

SUMMARY:
* Aphasia, the loss or impairment of language caused by brain damage, is one of the most devastating cognitive impairments of stroke. Aphasia can be treated with combination of speech-language therapy and drugs. Conventional speech-language therapy in chronic aphasic subjects is of little help and several drugs have been studied with limited success. Therefore other therapeutic strategies are warranted.
* Recent data suggest that drugs (memantine) acting on the brain chemical glutamate may help the recovery of cognitive deficits, included language, in subjects with vascular dementia. The present study examines the safety profile and efficacy of memantine paired with intensive language therapy in subjects with stroke-related chronic aphasia (more than 1 yr. of evolution).

DETAILED DESCRIPTION:
* The efficacy of drugs that act on glutamate such as the N-methyl-D-aspartic acid (NMDA) receptor antagonist memantine requires to be explored in this population. The rationale for using memantine in post-stroke aphasia comes from recent studies on vascular dementia. Data extracted from a recent Cochrane review of randomized controlled trials of memantine in different types of dementia (vascular dementia, Alzheimer's disease, mixed dementia) reveal, after 6 weeks of treatment, beneficial effects on cognition (including language), activities of daily living, behavior and global scales as well as in the global impression of change.
* Recovery from aphasia is possible even in severe cases. While speech-language therapy remains as the mainstay treatment of aphasia, its effectiveness has not been conclusively proved. This has motivated the planning of more rational therapies (e.g., constraint-induced language therapy [Pulvermüller et al., 2001; 32: 1621-1626]).
* In addition, the neural correlates of improvement of language function can now be readily detectable with event-related potentials. This is a noninvasive technique that can detect in real time functional brain changes during recovery promoted by the combined action of memantine and constraint-induced language therapy.
* The aim of the present study is to assess the efficacy, safety profile, and functional correlates of memantine paired with massed language therapy in a sample of patients with chronic poststroke aphasia.

ELIGIBILITY:
Inclusion Criteria:

* Chronic aphasia of more than one year duration
* Must be able to complete protocol

Exclusion Criteria:

* Dementia
* Major psychiatric illness
* Severe global aphasia (precludes participation in constraint-induced language therapy)

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2005-03; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Language function (overall aphasia severity). | 24 weeks

SECONDARY OUTCOMES:
Depression | 24 weeks
Cognitive evaluation of language function | 24 weeks
Changes in event-related potential | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo L. Berthier, M.D., Ph.D, Principal Investigator — Gabinete Berthier y Martínez and Centro de Investigaciones Médico-Sanitarias (CIMES), University of Malaga
Locations (1):
- Gabinete Berthier y Martínez and Centro de Investigaciones Médico-Sanitarias (CIMES) University of Malaga, Málaga, Malaga, Spain

REFERENCES:
- [Background] Orgogozo JM, Rigaud AS, Stoffler A, Mobius HJ, Forette F. Efficacy and safety of memantine in patients with mild to moderate vascular dementia: a randomized, placebo-controlled trial (MMM 300). Stroke. 2002 Jul;33(7):1834-9. doi: 10.1161/01.str.0000020094.08790.49. PMID 12105362
- [Background] Pantoni L. Treatment of vascular dementia: evidence from trials with non-cholinergic drugs. J Neurol Sci. 2004 Nov 15;226(1-2):67-70. doi: 10.1016/j.jns.2004.09.014. PMID 15537523
- [Background] Roman G. Perspectives in the treatment of vascular dementia. Drugs Today (Barc). 2000 Sep;36(9):641-53. doi: 10.1358/dot.2000.36.9.593781. PMID 12847569